CLINICAL TRIAL: NCT03133026
Title: The Role of Cholangioscopy and Biliary Radio Frequency Ablation in the Management of Occluded Biliary Self-expanding Metal Stent.
Brief Title: Cholangioscopic Assessment of Occluded Biliary Stent and Role of Biliary Radiofrequency Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AIG-001
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Jaundice; Cholangitis
Keywords: obstructive Jaundice; Self Expandable Metal Stents (SEMS); Cholangitis
MeSH Terms: conditions — Jaundice, Obstructive; Cholangitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sludge group (Active Comparator): If Single operator cholangioscopy reveals only sludge then sludge will be cleared using conventional technique during ERCP.
  Interventions: Device: Single operator cholangioscopy, Endoscopic biliary RFA
- Ingrowth / Overgrowth (Active Comparator): If Single operator cholangioscopy reveals tumour ingrowth or overgrowth then to evaluate the role of biliary RFA for occluded stent due to tumour ingrowth or overgrowth
  Interventions: Device: Single operator cholangioscopy, Endoscopic biliary RFA

INTERVENTIONS:
Device: Single operator cholangioscopy, Endoscopic biliary RFA — Single operator cholangioscopy will be done to acess the cause of occluded SEMS, if tumour ingrowth or overgrowth seen then endoscopic biliary RFA will be done
  Other Names: SpyGlass cholangioscopy

SUMMARY:
Primary Objective: To document state-of- the-art multi-modality management of occluded biliary SEMS aiming to minimize number of reinterventions while providing symptom relief without procedure-related serious adverse events.

NOTE: This study will be hypothesis-generating for an anticipated randomized controlled study (RCT) to compare outcomes of placement of a plastic stent inside the occluded SEMS to outcomes of the proposed multi-modality approach.

DETAILED DESCRIPTION:
Study Design:

Prospective, multi-center, single arm, post market, observational study

Two groups:

* Sludge group: SEMS occluded due to sludge/stones in SEMS
* Ingrowth/overgrowth group: SEMS occluded due to malignant tumor ingrowth or benign hyperplastic tissue overgrowth

Primary Endpoint:

Successful restoration of bile duct drainage with biliary obstructive symptom and cholangitis relief as applicable, without procedure related SAE'S, from procedure through 30 days of follow-up.

Secondary Endpoints:

1. Occurrence and severity of procedure related serious adverse events from procedure through 30 days after procedure
2. Resolution of cholangitis where applicable
3. Technical success of procedure performed for restoration of bile duct drainage, overall and stratified by treatment group Sludge group: Ability to restore stent patency by cleaning the stent content followed by cholangiographically or cholangioscopically confirmed restored stent patency Ingrowth / overgrowth group: Ability to perform biliary radio frequency ablation (RFA) followed by cholangiographically or cholangioscopically confirmed restored stent patency
4. Improvement of biliary obstructive symptoms at 1 week and 1 month post procedure compared to Baseline
5. Improvement of Laboratory Liver Function Tests (LFT) at 1 week and 1 month post procedure compared to Baseline
6. Biliary Reintervention rate from procedure through 30 days after procedure, including reinterventions caused by plastic stent occlusion
7. Impact of cholangioscopy on current standard of care, which is to place a stent inside the occluded SEMS by

   * Avoiding placement of a second stent (plastic or metal)
   * Avoiding a repeat ERCP
   * Reducing associated cost

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 or older 2. Willing and able to comply with the study procedures and provide written informed consent to participate in the study 3. Recurrent biliary obstructive symptoms after biliary SEMS placement 4. Biliary SEMS occlusion.

Exclusion Criteria:

* 1. Contraindications for endoscopic techniques 2. Ongoing cholangitis. NOTE: In case a patient presents who meets the inclusion and exclusion criteria, but has cholangitis, then a naso-biliary drain (NBD) will be placed before the ERCP until the cholangitis resolves.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Successful restoration of bile duct drainage | 1 month
  Successful restoration of bile duct drainage with biliary obstructive symptom and cholangitis relief as applicable, without procedure related SAE'S, from procedure through 30 days followup.

SECONDARY OUTCOMES:
Resolution of cholangitis | 1 week and 1 month
  1. Occurrence and severity of procedure related serious adverse events from procedure through 30 days after procedure 2. Resolution of cholangitis where applicable 4. Improvement of biliary obstructive symptoms at 1 week and 1 month post procedure compared to Baseline 5. Improvement of Laboratory Liver Function Tests (LFTs) at 1 week and 1 month post procedure compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Ramchandani, MD DM, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No